CLINICAL TRIAL: NCT03137121
Title: Olanzapine for the Treatment of Chronic Nausea and/or Vomiting, Unrelated to Chemotherapy or Radiation, in Advanced Cancer Patient - A Pilot, Dose-Finding Trial
Brief Title: Olanzapine for the Treatment of Chronic Nausea and/or Vomiting in Advanced Cancer Patients
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Collaborators: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Rudolph Navari, Professor, University of Alabama at Birmingham
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: F170104006 (XUAB 16100); 000515449 (Other: UAB Office of Sponsored Programs)
Record Dates: First submitted 2017-04-25; First posted 2017-05-02 (Actual); Results first posted 2021-08-17 (Actual); Last update posted 2021-08-17 (Actual); Status verified 2021-07

CONDITIONS: Advanced Cancer
Keywords: nausea; vomiting; olanzapine
MeSH Terms: conditions — Nausea; Vomiting | interventions — Olanzapine

STUDY DESIGN:
Intervention Model Description: There will be two groups for the study: Olanzapine Group will receive the study drug and Placebo Group will receive a placebo.
Who Masked: Participant, Care Provider, Investigator
Masking Description: Patients will receive the study drug or placebo in a double-blind fashion.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Olanzapine (Experimental): Patients will receive 5 mg olanzapine orally for 1 to 7 days daily.
  Interventions: Drug: Olanzapine
- Placebo (Placebo Comparator): Patients will receive a placebo orally for 1 to 7 days daily.
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Olanzapine — Olanzapine is used as an anti-emetic.
  Other Names: Zyprexa
  Arms: Olanzapine
Other: Placebo — The placebo is a non-anti-emetic.
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate the use of olanzapine for the treatment of cancer patients with chronic nausea and/or vomiting unrelated to chemotherapy or radiation in a randomized placebo-controlled pilot trial.

DETAILED DESCRIPTION:
Patients with advanced cancer experience a variety of physical and psychosocial symptoms that significantly affect the patients' quality of life. Chronic nausea is a particularly distressing symptom present in >60% of patients with advanced cancer. A number of palliative care studies have evaluated treatments of nausea with limited success. Olanzapine with its unique formulation and decreased drug interactions compared to many other drugs appears to be a reasonable candidate for further evaluation. Olanzapine has significant potential for use in the prevention and treatment of nausea in a palliative care setting with a once-daily dosing.

ELIGIBILITY:
Inclusion Criteria:

* Be at least 18 years of age
* Have histologically or cytologically-confirmed malignant disease in an advanced incurable stage
* Have not received chemotherapy or radiation for >14 days (advanced cancer patients receiving hormonal therapy or targeted therapy that does not come with a recommendation for prophylactic anti-emetic therapy are eligible)
* Have chronic nausea that has been present for at least one week (worst daily score >3, 0-10 visual analogue scale) or vomiting at least five times over past one week
* Have serum creatinine < 2.0 mg/dl and serum glutamic oxaloacetic transaminase (SGOT) or serum glutamic pyruvic transaminase (SGPT) < 3 times upper limits of normal ≤120 days prior to registration
* Absolute neutrophil count (ANC) >1500 mm3 <120 days prior to registration
* Women of childbearing potential must consent to use adequate contraception throughout protocol therapy; females of childbearing potential must have a negative urine pregnancy test <7 days prior to registration.

Exclusion Criteria:

* Not be receiving treatment with another antipsychotic agent such as risperidone, quetiapine, clozapine, phenothiazine or butyrophenone for less than or equal to 30 days prior to registration or planned during protocol therapy (patients may have received prochlorperazine and other phenothiazines as prior anti-emetic therapy)
* Not have concurrent use of ethyol
* Not have severe cognitive compromise
* History of central nervous system (CNS) disease (e.g. brain metastases, seizure disorder)
* Concurrent use of amifostine, concurrent abdominal radiotherapy; concurrent use of quinolone antibiotic therapy
* Chronic alcoholism (as determined by the investigator)
* Known hypersensitivity to olanzapine
* Known cardiac arrhythmia, uncontrolled congestive heart failure or acute myocardial infarction within the previous six months
* History of uncontrolled diabetes mellitus (stable insulin dose and/or stable oral hypoglycemic agent permitted)
* Planned chemotherapy or radiation during the 7 days following study initiation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2017-07-12 (Actual); Primary Completion 2019-07-12 (Actual); Study Completion 2020-09-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Rudolph Navari, MD, Principal Investigator — University of Alabama at Birmingham
Locations (5):
- United States (5):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Indiana University, Indianapolis, Indiana
  - Mayo Clinic, Rochester, Minnesota
  - Washington University School of Medicine, St Louis, Missouri
  - Hospital Sisters Health System (HSHS) St. Vincent Hospital, Green Bay, Wisconsin

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Navari RM, Pywell CM, Le-Rademacher JG, White P, Dodge AB, Albany C, Loprinzi CL. Olanzapine for the Treatment of Advanced Cancer-Related Chronic Nausea and/or Vomiting: A Randomized Pilot Trial. JAMA Oncol. 2020 Jun 1;6(6):895-899. doi: 10.1001/jamaoncol.2020.1052. PMID 32379269

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Olanzapine | Placebo
Started | 15 | 15
Completed | 15 | 14
Not Completed | 0 | 1
Not completed — Withdrawal by Subject | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Olanzapine | Placebo | Total
Number analyzed (Participants) | 15 | 15 | 30
Age, Continuous [Mean (Standard Deviation); unit: years] | 63 (9) | 60 (11) | 62 (7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 9 | 17
  Male | 7 | 6 | 13
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 15 | 15 | 30
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 5 | 6 | 11
  White | 10 | 9 | 19
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 15 | 15 | 30

OUTCOME MEASURES:

1. Primary Outcome: Mean Nausea Scores
Description: Daily nausea scores (the primary objective) on day 1 to 7 of treatment for each patient from the Olanzapine and Placebo group will be measured using the Visual Analogue Scale rankings from 0-10 where 0 is no nausea and 10 is the maximum nausea experienced by a patient. A Visual Analogue Scale is a psychometric response scale which can be used in questionnaires. It is a measurement instrument for subjective characteristics or attitudes that can't be directly measured.
  Patients will be asked to record the average nausea score for each day in a diary and a study nurse will call the patient at the same time each day to remind the patient to record the nausea score and to inquire about any toxicities. The difference in the nausea scores for the patients in each group (Olanzapine and Placebo) will be compared.
Time Frame: Nausea score from the Visual Analogue Scale will be recorded each day daily for 7 days. An average value calculated will be reported for the 7 day period.
Population: One patient withdrew on their own from the Placebo Group
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Olanzapine | Placebo
Number analyzed (Participants) | 15 | 14
units on a scale | 1 (1) | 9 (2)

2. Secondary Outcome: Number of Emetic Episodes
Description: The number of emetic episodes (a secondary outcome) by each patient in each group, Olanzapine & Placebo, on each day of treatment will be recorded by each patient on each day of treatment in a diary. A study nurse will contact each patient at the same time of each day of the study to ask the patient to record the number of emetic episodes and report any toxicities.The number of emetic episodes for the patients in each Group for each day of the treatment will be compared.
Time Frame: Number of emetic episodes for each patient on each day of the seven day treatment.
Population: One patient withdrew from the Placebo Group.
Measure: Number; unit: episodes
Arm/Group | Olanzapine | Placebo
Number analyzed (Participants) | 15 | 14
episodes
  day 1 | 3 | 3
  day 2 | 0 | 3
  day 3 | 0 | 3
  day 4 | 0 | 3
  day 5 | 0 | 3
  day 6 | 0 | 3
  day 7 | 0 | 3

3. Secondary Outcome: Number of Treatment-related Adverse Events as Assessed by CTCAE v4.0".
Description: Adverse events will be measured by patient-reported outcomes questionnaires and the Common Terminology Criteria for Adverse Events (CTCAE v4.0). A study nurse will contact each patient each day of the seven days of treatment to inquire about any toxicities, specifically sedation and appetite. Sedation and appetite will be reported by the patient in each Group on a Visual Analogue Scale of 0 to 10 with 0 being no sedation or no appetite to 10 indicating maximum sedation or maximum appetite.
Time Frame: Daily assessment for 7 days for each patient in Olanzapine & Placebo Groups.
Population: One patient withdrew from Placebo Group.
Measure: Number; unit: Events
Arm/Group | Olanzapine | Placebo
Number analyzed (Participants) | 15 | 14
Events | 3 | 21

ADVERSE EVENTS:
Time Frame: from baseline through 8 days
Description: One patient withdrew from Placebo Group.
Arm/Group | Olanzapine | Placebo
All-Cause Mortality (participants affected / at risk) | 0/15 | 0/14
Serious Adverse Events (participants affected / at risk) | 0/15 | 0/14
Other Adverse Events (participants affected / at risk) | 3/15 | 6/14
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Olanzapine (N=15) | Placebo (N=14)
Nausea (Gastrointestinal disorders) | 3 (3) | 6 (21)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-04-03): https://cdn.clinicaltrials.gov/large-docs/21/NCT03137121/Prot_SAP_000.pdf